CLINICAL TRIAL: NCT01753128
Title: Efficacy of Imipramine for Treatment of Patients With Esophageal
Brief Title: Efficacy of Imipramine for Treatment of Patients With Esophageal Hypersensitivity/ Functional Heartburn
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 334/2553 (EC3)
Record Dates: First submitted 2012-12-17; First posted 2012-12-20 (Estimated); Last update posted 2014-08-18 (Estimated); Status verified 2014-08

CONDITIONS: Gastroesophageal Reflux Disease
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Imipramine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- imipramine (Active Comparator)
  Interventions: Drug: imipramine

INTERVENTIONS:
Drug: imipramine

SUMMARY:
Esophageal hypersensitivity/Functional heartburn are common among non-erosive reflux disease (NERD) patients who do not response to proton pump inhibitors. Whether tricyclic antidepressant improves NERD patient's symptoms remains unknown

Aim of this randomized controlled trial study is to determine the efficacy of imipramine, which could increase esophageal pain thresholds in healthy volunteers, in comparison with placebo for treatment patients with esophageal hypersensitivity or functional heartburn evaluated by improvement of specific-symptom score and quality of life

ELIGIBILITY:
Inclusion Criteria:

* patient with typical reflux symptoms (heartburn and/or regurgitation) more than 3 times per week in at least last 3 months
* Age more than 18 years
* Upper GI endoscopy showed no esophageal mucosal breaks
* MII-pH monitoring was not showed abnormal both acid and non-acid reflux
* symptoms was not improved after received standard dose proton pump inhibitor for at least 1 month

Exclusion Criteria:

* history of thoracic, esophagus, or stomach surgery
* severe esophageal motility disorder eg. Achalasia, scleroderma, autonomic/peripheral neuropathy/myopathy
* patient who was indicated to receive proton pump inhibitor
* pregnant women
* patient who was allergy to imipramine
* patient who received tricyclic antidepressant or SSRI with in 3 month of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2012-12; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
improvement of GERD score | 6 months

SECONDARY OUTCOMES:
improve quality of life | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Julajak Limsrivilai, MD, Principal Investigator — Mahidol University
Locations (1):
- Medical Institue; Siriraj Hospital, Bangkok, Bangkok, Thailand